CLINICAL TRIAL: NCT05178498
Title: Longitudinal Study Evaluating the Impact of Dietary Inflammatory Potential on Breast Cancer Risk in a Cohort of Women Followed in the Breast Cancer Prevention Clinic at the Ohio State University Comprehensive Cancer Center- James Cancer Hospital and Solove Research Institute
Brief Title: Impact of Dietary Inflammatory Potential on Breast Cancer Risk
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sagar Sardesai, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-21065; NCI-2021-03342 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Atypical Ductal Hyperplasia; Breast Atypical Lobular Hyperplasia; Breast Carcinoma; Breast Lobular Carcinoma In Situ; Breast Sclerosing Adenosis
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Breast Carcinoma In Situ | interventions — Chromatin Immunoprecipitation Sequencing; Follow-Up Studies; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (physical exam, questionnaire): Patients complete physical measurements every 6 months and complete questionnaires annually for 5 years. Patients are followed up annually in years 5-10.
  Interventions: Procedure: Follow-Up; Procedure: Physical Examination; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Follow-Up — Undergo follow up
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
Procedure: Physical Examination — Complete physical measurements
  Other Names: Assessment; General Examination; Physical; Physical Assessment; Physical Exam; physical_exam
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study evaluates the association of dietary inflammatory potential with breast cancer risk. Information collected in this study may help doctors to identify modifiable risk factors, screen high risk patients early, improve prevention strategies, and provide timely intervention for early therapeutic management as needed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the association of dietary inflammatory potential (measured by Empirical Dietary Inflammatory Pattern [EDIP] score) at baseline using Diet History Questionnaire III (DHQIII) food frequency questionnaire (FFQ) with the incidence of breast cancer in high risk women established in the breast cancer prevention clinic at Ohio State University Comprehensive Cancer Center (OSUCCC) - James.

SECONDARY OBJECTIVES:

I. To evaluate changes in inflammatory potential of diet (EDIP score) from baseline FFQ and subsequently administered annually, and determine how these dietary changes relate to breast cancer risk longitudinally.

II. To evaluate associations of dietary inflammatory potential (EDIP score) with measures of obesity including bone marrow index (BMI) (obesity defined as >= 30, non-obese < 30) and abdominal/visceral adiposity (waist-hip ratio [WHR] > 0.85 or waist circumference [WC] >= 80 cm in women) at baseline.

III. To evaluate the association of dietary inflammatory potential (EDIP score) with mammographic breast density by breast imaging reporting and data system (BIRADS) classification at baseline.

CORRELATIVE OBJECTIVES:

I. To evaluate the correlation of baseline and annual inflammatory blood-based biomarkers (IL-6, hsCRP, adiponectin, leptin, insulin resistance [Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)]) with: a) dietary inflammatory potential (EDIP score) and b) visceral adiposity (waist-hip ratio > 0.85 or waist circumference >= 80 cm in women) and c) mammographic breast density by BIRADS classification at baseline and longitudinally (every year for 5 years).

II. To evaluate the association of baseline circulating biomarkers (hsCRP, TNF-a, insulin resistance [HOMA-IR]) and breast cancer incidence longitudinally in high risk patients.

EXPLORATORY OBJECTIVES:

I. Describe utilization of supplemental imaging by type, including breast magnetic resonance imaging (MRI), automated breast ultrasound (ABUS) and contrasted-enhanced spectral mammography (CESM), in all enrolled women.

II. Describe use of chemoprevention strategies (initiation of tamoxifen, raloxifene, aromatase inhibitor (AI), or other) in women presenting at the high risk clinic at OSUCCC-James.

OUTLINE:

Patients complete physical measurements every 6 months and complete questionnaires annually for 5 years. Patients are followed up annually in years 5-10.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Established in the high risk clinic at OSUCCC- James (includes patients with family history of breast cancer [BC], known genetic predisposition, personal history of known atypia/breast lobular carcinoma in situ [LCIS], or prior chest wall radiation)
* Patients at high risk for BC established in the surgical oncology clinic at Stefanie Spielman Comprehensive Breast Center (SSCBC), with one of the following diagnoses: Atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH), lobular carcinoma in situ (LCIS), sclerosing adenosis (SA), or radial scars (RS)
* Able to read and understand English
* Able to provide informed consent
* Must consent to continued follow-up of medical records during the study period

Exclusion Criteria:

* Prisoners
* Not able to speak and understand English
* Known personal history of ductal carcinoma in situ (DCIS) or Invasive BC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to breast cancer events during study follow up | Up to 10 years
  Will be expressed as the means, medians and standard deviations (for continuous variables) or frequencies and percentages (for categorical variables). To assess the association of baseline Empirical Dietary Inflammatory pattern (EDIP) scores with breast cancer incidence, Cox proportional hazards regression will be used to estimate the hazard ratio (HR) and its 95% confidence interval (CI).

SECONDARY OUTCOMES:
Bone marrow index | Up to 10 years
  Will be expressed as the means, medians and standard deviations (for continuous variables) or frequencies and percentages (for categorical variables).
Waist-hip ratio | Up to 10 years
  Will be expressed as the means, medians and standard deviations (for continuous variables) or frequencies and percentages (for categorical variables).
Waist circumference | Up to 10 years
  Will be expressed as the means, medians and standard deviations (for continuous variables) or frequencies and percentages (for categorical variables).
Mammographic breast density | Up to 10 years
  Will be measured by breast imaging reporting and data system. Will be expressed as the means, medians and standard deviations (for continuous variables) or frequencies and percentages (for categorical variables).

OTHER OUTCOMES:
Proportion of patients who received at least 1 supplemental screening breast by breast magnetic resonance imaging, automated breast ultrasound, and contrasted-enhanced spectral mammography during study follow up | Up to 12 months
Proportion of patients initiating chemoprevention during study follow up | Up to 12 months
  Proportion of patients initiating chemoprevention within 12 months of enrollment will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar D Sardesai, MSPH, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu